CLINICAL TRIAL: NCT02169401
Title: a PRospEctive Post Market Trial of Drg stImulation With the Commercially Available Axium
Brief Title: A Multi-centre Observational Study of the Axium Neurostimulator as a Treatment for Chronic Pain
Acronym: PREDICT
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 08-SMI-2012 - PREDICT
Record Dates: First submitted 2014-06-13; First posted 2014-06-23 (Estimated); Results first posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-09

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Treated subjects: All subjects recruited and treated with the Axium Neurostimulator
  Interventions: Device: Implantation with the commercially available Axium Neurostimulator

INTERVENTIONS:
Device: Implantation with the commercially available Axium Neurostimulator

SUMMARY:
08-SMI-2012 is a post market, observational, questionnaire based study to assess the effectiveness of the commercially available Axium neurostimulator in the management of intractable, chronic pain.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years old
2. Subject is able and willing to comply with the follow-up schedule and protocol
3. Chronic, intractable pain for at least 6 months
4. Failed conservative treatments for chronic pain including but not limited to pharmacological therapy, physical therapy and interventional pain procedures for chronic pain
5. Average baseline pain rating of 60 mm on the Visual Analog Scale in the primary region of pain
6. In the opinion of the Investigator, the subject is psychologically appropriate for the implantation for an active implantable medical device
7. Subject is able to provide written informed consent

Exclusion Criteria:

1. Female subject of childbearing potential is pregnant/nursing, plans to become pregnant or is unwilling to use approved birth control
2. Escalating or changing pain condition within the past month as evidenced by investigator examination
3. Subject has had corticosteroid therapy at an intended site of stimulation within the past 30 days
4. Subject has had radiofrequency treatment of an intended target DRG within the past 3 months
5. Subject currently has an active implantable device including implantable cardioverter defibrillator, pacemaker, spinal cord stimulator or intrathecal drug pump
6. Subject is unable to operate the device
7. Subjects currently has an active infection
8. Subject has, in the opinion of the Investigator, a medical comorbidity that contraindicates placement of an active medical device
9. Subject has participated in another clinical trial within 30 days
10. Subject has a coagulation disorder or uses anticoagulants that, in the opinion of the investigator, precludes participation
11. Subject has been diagnosed with cancer in the past 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic Pain Patients
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2012-11; Primary Completion 2017-01-25 (Actual); Study Completion 2017-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: S ElDabe, Prof, Principal Investigator — James Cook University Hospital
Locations (1):
- James Cook University Hospital, Middlesbrough, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Treated Subjects: All subjects recruited and treated with the Axium Neurostimulator.
  Implantation with the commercially available Axium Neurostimulator.
Period: Overall Study
Arm/Group | Treated Subjects
Started | 135
Completed | 108
Not Completed | 27

BASELINE CHARACTERISTICS:
Arm/Group | Treated Subjects
Number analyzed (Participants) | 135
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 122
  >=65 years | 13
Age, Continuous [Mean (Full Range); unit: years] | 49 [22 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 77
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: 3 subjects did not disclose their race
  Participants
    Race: number analyzed (Participants) | 132
    Race: Caucasian/White | 130
    Race: Asian | 1
    Race: Afro-Caribbean | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 135
Weight [Mean (Full Range); unit: kg] — Population: Weight was not available for 7 subjects.
  kg
    number analyzed (Participants) | 128
    (all) | 81 [47 to 135]
Height [Mean (Full Range); unit: cm] — Population: Height not available for 2 subjects.
  cm
    number analyzed (Participants) | 133
    (all) | 160 [148 to 195]

OUTCOME MEASURES:

1. Primary Outcome: Pain Relief- Change in VAS Pain Intensity From Baseline to Post Implantation
Description: The visual analog is a widely accepted measure of pain intensity. VAS scale ranges from 0 to 10, where 0 is the minimum and 10 is the maximum score. A higher score indicates greater pain intensity (listed below are some citations to illustrate this point). An increase in VAS scores conveys an increase in pain.
  Jensen, Mark P., Connie Chen, and Andrew M. Brugger. "Interpretation of visual analog scale ratings and change scores: a reanalysis of two clinical trials of postoperative pain." The Journal of pain 4.7 (2003): 407-414. MPQ, M. (2011). Measures of adult pain. Arthritis Care Res., 63, S240-S252. Hawker, G. A., Mian, S., Kendzerska, T., & French, M. (2011). Measures of adult pain: Visual analog scale for pain (vas pain), numeric rating scale for pain (nrs pain), mcgill pain questionnaire (mpq), short-form mcgill pain questionnaire (sf-mpq), chronic pain grade scale (cpgs), short form-36 bodily pain scale (sf-36 bps), and measure of intermittent and constant osteoarthritis pain.
Time Frame: Post implantation at; 1, 3, 6, 12 and 24 months
Population: Subject attrition reduced the number of participating and analyzable subjects at all subsequent visits post-implant.
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Treated Subjects: All subjects who receive the Axium neurostimulator
Arm/Group | Treated Subjects
Number analyzed (Participants) | 135
cm
  Baseline: number analyzed (Participants) | 133
  Baseline | 7.5 (1.7)
  1-Month Visit: number analyzed (Participants) | 98
  1-Month Visit | 4.4 (2.8)
  3-Month Visit: number analyzed (Participants) | 95
  3-Month Visit | 5.2 (2.5)
  6-Month Visit: number analyzed (Participants) | 90
  6-Month Visit | 4.7 (2.6)
  12-Month Visit: number analyzed (Participants) | 83
  12-Month Visit | 4.9 (2.8)
  24-Month Visit: number analyzed (Participants) | 73
  24-Month Visit | 4.4 (2.8)

ADVERSE EVENTS:
Time Frame: Adverse Event data collected from the time subject is enrolled (upon informed consent) through 6 months follow-up or withdrawal, whichever occurred first.
Description: Adverse Event - untoward medical occurrence, unintended disease/injury, untoward clinical sign whether or not related to the investigational device. Serious criteria: AE that led to death, serious deterioration subject health or fetal distress, death or congenital abnormality/birth defect.
Groups:
- Treated Subjects: All subjects treated with the Axium Neurostimulator.
Arm/Group | Treated Subjects
All-Cause Mortality (participants affected / at risk) | 2/135
Serious Adverse Events (participants affected / at risk) | 4/135
Other Adverse Events (participants affected / at risk) | 35/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated Subjects (N=135)
Pain/discomfort in target area (General disorders) | 1 (1)
Abcess at lead site (Skin and subcutaneous tissue disorders) | 1 (1)
Leg pain and numbness (General disorders) | 1 (1)
Loss of stimulation (Product Issues) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated Subjects (N=135)
Pain/discomfort at IPG site (General disorders) | 15 (15)
Lead migration (Product Issues) | 7 (7)
IPG migration (Product Issues) | 2 (2)
Increasing pain in target area (General disorders) | 1 (1)
Painful/unpleasant stimulation (General disorders) | 2 (2)
Pain/discomfort at IPG site and pain in leg (General disorders) | 1 (1)
Cerebral spinal fluid leakage (Surgical and medical procedures) | 1 (1)
Lead impedance out of range (Product Issues) | 1 (1)
Skin erosion (Skin and subcutaneous tissue disorders) | 1 (1)
Foreign object in epidural space (Musculoskeletal and connective tissue disorders) | 1 (1)
Loss of stimulation (Product Issues) | 3 (3)
Pocket infection (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol (2014-03-13): https://cdn.clinicaltrials.gov/large-docs/01/NCT02169401/Prot_000.pdf